CLINICAL TRIAL: NCT04379427
Title: Measurement Algorithm Control and Optimization With Subsequent Performance Evaluation of Sanmina Non-invasive Biosensors During a Standardized Meal Test in Patients With Diabetes Mellitus Type 1 and Type 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sciema UG (Other)
Collaborators: Sanmina (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: SNM-NGM-001
Record Dates: First submitted 2020-04-29; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The first 2 study parts include 12 patients each. In the third study part 36 patients will be enrolled. Study part 1 and 2 will be used for optimization and control of the measurement algorithms of the Sanmina biosensors. During the third study part with enrolment of 36 patients, the precision and accuracy of the final Sanmina biosensor algorithm will be demonstrated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Optimization and control 1 (Experimental): The first study part/arm includes 12 patients and will be used for optimization and control of the measurement algorithms of the Sanmina biosensors.
  Interventions: Device: Sanmina Biosensor
- Optimization and control 2 (Experimental): The second study part/arm includes 12 patients and will be used for optimization and control of the measurement algorithms of the Sanmina biosensors.
  Interventions: Device: Sanmina Biosensor
- Precision and accuracy (Other): During the third study part with enrolment of 36 patients, the precision and accuracy of the final Sanmina biosensor algorithm will be demonstrated.
  Interventions: Device: Sanmina Biosensor

INTERVENTIONS:
Device: Sanmina Biosensor — non-invasive blood glucose measurement using the Sanmina Biosensor referenced with the invasive reference blood glucose device YSI 2400 Plus.

SUMMARY:
Measurement algorithm control and optimization with subsequent performance evaluation of Sanmina biosensors in monitoring of glucose, heart rate (HR), and SpO2 in patients with type 1 and type 2 diabetes during a standardized meal experiment.

DETAILED DESCRIPTION:
* This study is a combined, open label, prospective, comparative single-center study.
* The study is separated in 3 consecutive study parts. The first 2 study parts include 12 patients each. In the third study part 36 patients will be enrolled. Study part 1 and 2 will be used for optimization and control of the measurement algorithms of the Sanmina biosensors. During the third study part with enrolment of 36 patients, the precision and accuracy of the final Sanmina biosensor algorithm will be demonstrated. The study conduct for all 60 participants of all 3 study parts will be exactly the same. In all groups of participants, the Sanmina finger clip and wearable non-invasive monitoring biosensor will be individually introduced and assigned. During the study visit at the study site, a standardized meal will be given to the participants. At eleven time points before and after the standardized meal, glucose, heart rate, and pO2 will be measured using the Sanmina finger clip and wearable non-invasive monitoring biosensor. The measurement time points are -30, 0, 15, 30, 45, 60, 75, 90, 120, 150 and 180 min. The measurements will be compared to capillary blood glucose measurements by YSI Stat 2300 and StatStrip (glucose), and parallel measurements of the heart rate and the pO2 using a patient monitor. Further the exact skin colour will be evaluated using a skin colour card.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetic subjects or healthy probands
* Subjects who are able to complete informed consent form (by him/herself or by his/her guardian);
* 18 years old and above;
* Anatomically suitable finger in discretion of the investigator

Exclusion Criteria:

* Does not meet inclusion criteria;
* Any conditions that may hamper good visual contact between the finger or wrist and sensor, such as raised birthmarks, scars, tattoos;
* Pregnancy;
* Nursing mothers;
* Any skin scratch(es), damage, over dry, long nails on the measured finger;
* Unsuitable finger with the device might be excluded if recognized during the trial;
* Medication containing nitrates

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Performance and accuracy of glucose levels | approx. 240 minutes
  performance and accuracy of the Sanmina biosensors (wearable and finger clip) in monitoring glucose levels (mg/dL) during a standardized meal experiment. Measurements (during the meal experiment) of the Sanmina biosensor will be compared to the capillary blood glucose reference method YSI STAT 2300 (glucose, in mg/dL).
Performance and accuracy of pO2 | approx. 240 minutes
  performance and accuracy of the Sanmina biosensors (wearable and finger clip) in monitoring pO2 (%) during a standardized meal experiment. PO2-measurements (during the meal experiment) of the Sanmina biosensor will be compared to the patient monitor (%).
Performance and accuracy of heart rate | approx. 240 minutes
  performance and accuracy of the Sanmina biosensors (wearable and finger clip) in monitoring heart rate (pulse/min) during a standardized meal experiment. Heart rate measurements (during the meal experiment) of the Sanmina biosensor will be compared to the patient monitor heart rate(pulse/min).

CONTACTS AND LOCATIONS:
Locations (1):
- Pfuetzner Science & Health Institute GmbH, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No